CLINICAL TRIAL: NCT06345586
Title: Drospirenone Only Pills and Cervical Mucus Changes in Obese Thai Women: A Pre- and Post-Bariatric Surgery Study
Brief Title: Drospirenone Only Pills and Cervical Mucus Changes: A Pre- and Post-Bariatric Surgery Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 078066
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-03

CONDITIONS: Contraception
Keywords: Drospirenone only pills; Obesity; Bariatric surgery; Roux-en-Y gastric bypass; Cervical mucus
MeSH Terms: conditions — Obesity | interventions — drospirenone

STUDY DESIGN:
Intervention Model Description: Participants received Drospirenone will be assess for cervical mucus change by modified Insler score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drospirenone (Experimental): Participants received Drospirenone 4 mg tablet orally once daily for 21-28 days
  Interventions: Drug: Drospirenone

INTERVENTIONS:
Drug: Drospirenone — 4 mg tablet once daily

SUMMARY:
The purpose of this study is to study the effect of Drospirenone on cervical mucus change by modified Insler score, pre-bariatric surgery and post-bariatric surgery

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent who meet the eligibility requirements will take Drospirenone-only pills (4 mg, once daily). Cervical mucus by modified Insler score will be evaluated on Day 4-7 of Drospirenone taking. Pre-bariatric surgery results will be compared with post-bariatric surgery results.

ELIGIBILITY:
Inclusion Criteria:

* Thai women aged 18-45 years who are obese and had an appointment for Bariatric surgery at Chulalongkorn Hospital
* Need contraception
* Able to use non-hormonal contraception during the study
* Giving consent

Exclusion Criteria:

* Pregnancy or history of giving birth within 3 months
* Breastfeeding within the 6 months
* History of using DMPA within 12 months
* History of using other types of hormonal birth control pills within 4 weeks
* History of bilateral oophorectomy or hysterectomy
* Suspected ovarian tumor or pathological ovarian cyst
* Regular cigarette smoking
* Contraindications to Drospirenone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Cervical mucus by modified Insler score | 1 month before and 1 month after bariatric surgery
  Modified Insler score (ferning, spinnbarkeit, viscosity, cellularity) according to the World Health Organization (WHO) guidelines 2010 used for prediction and detection of ovulation.
  Score ≥9 favoring fertility, 5-8 intermediate, and ≤4 unfavorable to fertility Comparing pre-bariatric surgery with post-bariatric surgery

SECONDARY OUTCOMES:
Estrogen and progesterone levels versus time | 1 month before and 1 month after bariatric surgery
  Serum estrogen and progesterone levels will be measured to evaluate change over time (pattern and value) and assess ovulation
Number of Participants With Treatment-Related Adverse Events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Punyawee Utaipatanacheep, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Currently have no recruited participant.

REFERENCES:
- [Result] Techagumpuch A, Pantanakul S, Chansaenroj P, Boonyagard N, Wittayapairoch J, Poonthananiwatkul T, et al. Thai Society for metabolic and bariatric surgery consensus guideline on bariatric surgery for the treatment of obese patient in Thailand. JAGST 2021;4:5-18.
- [Result] Simmons K, Edelman A. Contraception in the setting of obesity and bariatric surgery. In: Allen RH, Cwiak CA, editors. Contraception for the medically challenging patient. New York: Springer; 2014. P. 157-80.
- [Result] ACOG practice bulletin no. 105: bariatric surgery and pregnancy. Obstet Gynecol. 2009 Jun;113(6):1405-1413. doi: 10.1097/AOG.0b013e3181ac0544. No abstract available. PMID 19461456
- [Result] Ciangura C, Coupaye M, Deruelle P, Gascoin G, Calabrese D, Cosson E, Ducarme G, Gaborit B, Lelievre B, Mandelbrot L, Petrucciani N, Quilliot D, Ritz P, Robin G, Salle A, Gugenheim J, Nizard J; BARIA-MAT Group. Clinical Practice Guidelines for Childbearing Female Candidates for Bariatric Surgery, Pregnancy, and Post-partum Management After Bariatric Surgery. Obes Surg. 2019 Nov;29(11):3722-3734. doi: 10.1007/s11695-019-04093-y. PMID 31493139
- [Result] Mechanick JI, Apovian C, Brethauer S, Timothy Garvey W, Joffe AM, Kim J, Kushner RF, Lindquist R, Pessah-Pollack R, Seger J, Urman RD, Adams S, Cleek JB, Correa R, Figaro MK, Flanders K, Grams J, Hurley DL, Kothari S, Seger MV, Still CD. Clinical Practice Guidelines for the Perioperative Nutrition, Metabolic, and Nonsurgical Support of Patients Undergoing Bariatric Procedures - 2019 Update: Cosponsored by American Association of Clinical Endocrinologists/American College of Endocrinology, The Obesity Society, American Society for Metabolic and Bariatric Surgery, Obesity Medicine Association, and American Society of Anesthesiologists. Obesity (Silver Spring). 2020 Apr;28(4):O1-O58. doi: 10.1002/oby.22719. PMID 32202076
- [Result] Mengesha BM, Carter JT, Dehlendorf CE, Rodriguez AJ, Steinauer JE. Perioperative pregnancy interval, contraceptive counseling experiences, and contraceptive use in women undergoing bariatric surgery. Am J Obstet Gynecol. 2018 Jul;219(1):81.e1-81.e9. doi: 10.1016/j.ajog.2018.04.008. Epub 2018 Apr 7. PMID 29634911
- [Result] United Nations Department of Economic and Social Affairs, Population Division (2022). World Contraceptive Use 2022 [Internet]. [cited 9 August 2023]. Available from: https://www.un.org/development/desa/pd/data/world-contraceptive-use.
- [Result] Nightingale AL, Lawrenson RA, Simpson EL, Williams TJ, MacRae KD, Farmer RD. The effects of age, body mass index, smoking and general health on the risk of venous thromboembolism in users of combined oral contraceptives. Eur J Contracept Reprod Health Care. 2000 Dec;5(4):265-74. doi: 10.1080/13625180008500402. PMID 11245554
- [Result] Jick H, Jick SS, Gurewich V, Myers MW, Vasilakis C. Risk of idiopathic cardiovascular death and nonfatal venous thromboembolism in women using oral contraceptives with differing progestagen components. Lancet. 1995 Dec 16;346(8990):1589-93. doi: 10.1016/s0140-6736(95)91928-7. PMID 7500750
- [Result] Effect of different progestagens in low oestrogen oral contraceptives on venous thromboembolic disease. World Health Organization Collaborative Study of Cardiovascular Disease and Steroid Hormone Contraception. Lancet. 1995 Dec 16;346(8990):1582-8. PMID 7500749
- [Result] Rosano GMC, Rodriguez-Martinez MA, Spoletini I, Regidor PA. Obesity and contraceptive use: impact on cardiovascular risk. ESC Heart Fail. 2022 Dec;9(6):3761-3767. doi: 10.1002/ehf2.14104. Epub 2022 Sep 14. PMID 36103980
- [Result] Cardiovascular disease and use of oral and injectable progestogen-only contraceptives and combined injectable contraceptives. Results of an international, multicenter, case-control study. World Health Organization Collaborative Study of Cardiovascular Disease and Steroid Hormone Contraception. Contraception. 1998 May;57(5):315-24. PMID 9673838
- [Result] Vasilakis C, Jick H, del Mar Melero-Montes M. Risk of idiopathic venous thromboembolism in users of progestagens alone. Lancet. 1999 Nov 6;354(9190):1610-1. doi: 10.1016/S0140-6736(99)04394-9. PMID 10560680
- [Result] WHO Guidelines Approved by the Guidelines Review Committee. Medical Eligibility Criteria for Contraceptive Use. 5 ed. Geneva: World Health Organization Copyright © World Health Organization 2015.; 2015. p. 156-85.
- [Result] Curtis KM, Tepper NK, Jatlaoui TC, Berry-Bibee E, Horton LG, Zapata LB, Simmons KB, Pagano HP, Jamieson DJ, Whiteman MK. U.S. Medical Eligibility Criteria for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(3):1-103. doi: 10.15585/mmwr.rr6503a1. PMID 27467196
- [Result] Palacios S, Colli E, Regidor PA. Efficacy and cardiovascular safety of the new estrogen-free contraceptive pill containing 4 mg drospirenone alone in a 24/4 regime. BMC Womens Health. 2020 Oct 2;20(1):218. doi: 10.1186/s12905-020-01080-9. PMID 33008401
- [Result] Palacios S, Regidor PA, Colli E, Skouby SO, Apter D, Roemer T, Egarter C, Nappi RE, Skrivanek A, Jakimiuk AJ, Weyers S, Acs N, Elia D, Gemzell Danielsson K, Bitzer J. Oestrogen-free oral contraception with a 4 mg drospirenone-only pill: new data and a review of the literature. Eur J Contracept Reprod Health Care. 2020 Jun;25(3):221-227. doi: 10.1080/13625187.2020.1743828. Epub 2020 Apr 21. PMID 32312141
- [Result] Creinin MD, Angulo A, Colli E, Archer DF. The efficacy, safety, and tolerability of an estrogen-free oral contraceptive drospirenone 4 mg (24/4-day regimen) in obese users. Contraception. 2023 Dec;128:110136. doi: 10.1016/j.contraception.2023.110136. Epub 2023 Aug 5. PMID 37544572
- [Result] Archer DF, Ahrendt HJ, Drouin D. Drospirenone-only oral contraceptive: results from a multicenter noncomparative trial of efficacy, safety and tolerability. Contraception. 2015 Nov;92(5):439-44. doi: 10.1016/j.contraception.2015.07.014. Epub 2015 Jul 29. PMID 26232513
- [Result] Schlatter J. Oral Contraceptives after Bariatric Surgery. Obes Facts. 2017;10(2):118-126. doi: 10.1159/000449508. Epub 2017 Apr 22. PMID 28433989
- [Result] Krepelka P. New estrogen-free oral hormonal contraceptive (Estrogene free ill-EFP). Ceska Gynekol. 2020 Winter;85(3):222-225. PMID 33562977
- [Result] Duijkers IJ, Heger-Mahn D, Drouin D, Skouby S. A randomised study comparing the effect on ovarian activity of a progestogen-only pill (POP) containing desogestrel and a new POP containing drospirenone in a 24/4 regimen. Eur J Contracept Reprod Health Care. 2015;20(6):419-27. doi: 10.3109/13625187.2015.1044082. Epub 2015 Jun 15. PMID 26073333
- [Result] Han L, Creinin MD, Hemon A, Glasier A, Chen MJ, Edelman A. Mechanism of action of a 0.075 mg norgestrel progestogen-only pill 2. Effect on cervical mucus and theoretical risk of conception. Contraception. 2022 Aug;112:43-47. doi: 10.1016/j.contraception.2022.03.016. Epub 2022 Mar 31. PMID 35367204
- [Result] Moghissi KS, Marks C. Effects of microdose norgestrel on endogenous gonadotropic and steroid hormones, cervical mucus properties, vaginal cytology, and endometrium. Fertil Steril. 1971 Jul;22(7):424-34. doi: 10.1016/s0015-0282(16)38342-x. No abstract available. PMID 5104921
- [Result] FSRH Guideline (August 2022) Progestogen-only Pills. BMJ Sex Reprod Health. 2022 Aug;48(Suppl 1):1-75. doi: 10.1136/bmjsrh-2022-PoP. No abstract available. PMID 36316023
- [Result] Brache V, Cochon L, Duijkers IJ, Levy DP, Kapp N, Monteil C, Abitbol JL, Klipping C. A prospective, randomized, pharmacodynamic study of quick-starting a desogestrel progestin-only pill following ulipristal acetate for emergency contraception. Hum Reprod. 2015 Dec;30(12):2785-93. doi: 10.1093/humrep/dev241. Epub 2015 Sep 23. PMID 26405263
- [Result] Trevor G Cooper. WHO laboratory manual for the Examination and processing of human semen.5th ed. Switzerland: WHO; 2010. Appendix 5, Cervical mucus; p. 245-53.
- [Result] Tworoger SS, Hankinson SE. Collection, processing, and storage of biological samples in epidemiologic studies: sex hormones, carotenoids, inflammatory markers, and proteomics as examples. Cancer Epidemiol Biomarkers Prev. 2006 Sep;15(9):1578-81. doi: 10.1158/1055-9965.EPI-06-0629. PMID 16985015
- [Result] Taieb J, Benattar C, Birr AS, Lindenbaum A, Frydman R, Olivennes F. Delayed assessment of serum and whole blood estradiol, progesterone, follicle-stimulating hormone, and luteinizing hormone kept at room temperature or refrigerated. Fertil Steril. 2000 Nov;74(5):1053-4. doi: 10.1016/s0015-0282(00)01546-6. No abstract available. PMID 11056261
- [Result] Jane Ellis M, Livesey JH, Evans MJ. Hormone stability in human whole blood. Clin Biochem. 2003 Mar;36(2):109-12. doi: 10.1016/s0009-9120(02)00440-x. PMID 12633759
- [Result] Glasier A, Edelman A, Creinin MD, Han L, Matulich MC, Brache V, Westhoff CL, Hemon A. Mechanism of action of norgestrel 0.075 mg a progestogen-only pill. I. Effect on ovarian activity. Contraception. 2022 Aug;112:37-42. doi: 10.1016/j.contraception.2022.03.022. Epub 2022 Mar 26. PMID 35351445
- [Result] Wathen NC, Perry L, Lilford RJ, Chard T. Interpretation of single progesterone measurement in diagnosis of anovulation and defective luteal phase: observations on analysis of the normal range. Br Med J (Clin Res Ed). 1984 Jan 7;288(6410):7-9. doi: 10.1136/bmj.288.6410.7. PMID 6418326
- [Result] Landgren BM, Unden AL, Diczfalusy E. Hormonal profile of the cycle in 68 normally menstruating women. Acta Endocrinol (Copenh). 1980 May;94(1):89-98. doi: 10.1530/acta.0.0940089. No abstract available. PMID 6770571